CLINICAL TRIAL: NCT04472546
Title: Using the SpiderMass(TM) for in Vivo and Real Time Mass Spectrometry Analysis of Subject's Epidermis Suffering From Chronic Inflammatory Dermatosis Compared to Control Groups
Brief Title: Use of the SpiderMass for in Vivo Analysis of the Skin in Five Chronic Inflammatory Dermatosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SMPATHO01; 2019-A02105-52 (Other: ID-RCB)
Record Dates: First submitted 2020-06-05; First posted 2020-07-15 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Acne; Atopic Dermatitis; Psoriasis Vulgaris; Rosacea; Seborrheic Dermatitis; Healthy
Keywords: dermatitis; acne of the face; Atopic Dermatitis of the upper limb; Psoriasis Vulgaris; Rosacea; seborrheic dermatitis; SpiderMass; Lipid Index; Laser; Hydratation index; Transepidermal water loss; Scotch sampling; Absorbant paper
MeSH Terms: conditions — Acne Vulgaris; Dermatitis, Atopic; Rosacea; Dermatitis, Seborrheic; Dermatitis

STUDY DESIGN:
Intervention Model Description: Subject group :
  Exploratory study, monocentric and comparative performed at:
  * control subject group, divided in 5 subgroups :
    * A': associated to acne of the face subgroup
    * B' : associated to atopic dermatitis of the upper limb subgroup
    * C' : associated to vulgar plaque psoriasis subgroup
    * D' : associated to telangiectasic erythrocouperosis papule of the face (rosacea) subgroup
    * E' : associated to seborrheic dermatitis of scalp subgroup
  * subject group with dermatitis, divided in 5 subgroups :
    * A: acne of the face subgroup
    * B : atopic dermatitis of the upper limb subgroup
    * C : vulgar plaque psoriasis subgroup
    * D : telangiectasic erythrocouperosis papule of the face (rosacea) subgroup
    * E : seborrheic dermatitis of scalp subgroup
  Visit number :
  It includes 1 unique visit to the Skin Research Center, Toulouse, France. The maximum duration of participation for a subject is 1 day (around 2 hours).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control subject group (Other): Divided in 5 subgroups :
  * A': associated to acne of the face subgroup
  * B' : associated to atopic dermatitis of the upper limb subgroup
  * C' : associated to vulgar plaque psoriasis subgroup
  * D' : associated to telangiectasic erythrocouperosis papule of the face (rosacea) subgroup
  * E' : associated to seborrheic dermatitis of scalp subgroup
  Interventions: Other: in-vivo mesure; Other: Scotch; Other: Lipid index; Other: Absorbant paper; Other: Hydratation Index; Other: TransEpidermal Water Loss
- Subject group with dermatitis (Other): Divided in 5 subgroups :
  * A : acne of the face subgroup
  * B : Atopic dermatitis of the upper limb subgroup
  * C : Vulgar plaque psoriasis subgroup
  * D : Telangiectasic erythrocouperosis papule of the face (rosacea) subgroup
  * E : Seborrheic dermatitis of scalp subgroup
  Interventions: Other: in-vivo mesure; Other: Scotch; Other: Lipid index; Other: Absorbant paper; Other: Hydratation Index; Other: TransEpidermal Water Loss

INTERVENTIONS:
Other: in-vivo mesure — * for acne of the face subgroup and its associated control : face and inner side of the forearm
  * for atopic dermatitis of the upper limb subgroup and its associated control: upper limb (hand excluded) and inner side of the forearm
  * for vulgar plaque psoriasis subgroup and its associated control: upper limb (hand excluded) or lower limb and inner side of the forearm
  * for telangiectasic erythrocouperosis papule of the face (rosacea) subgroup and its associated control: face and inner side of the forearm
  * for seborrheic dermatitis of scalp subgroup and its associated control: scalp and inner side of the forearm
  Other Names: SpiderMass mesure
Other: Scotch — * for acne of the face subgroup and its associated control : face and inner side of the forearm
  * for atopic dermatitis of the upper limb subgroup and its associated control: upper limb (hand excluded) and inner side of the forearm
  * for vulgar plaque psoriasis subgroup and its associated control: upper limb (hand excluded) or lower limb and inner side of the forearm
  * for telangiectasic erythrocouperosis papule of the face (rosacea) subgroup and its associated control: face and inner side of the forearm
  * for seborrheic dermatitis of scalp subgroup and its associated control: scalp and inner side of the forearm
Other: Lipid index — * for acne of the face subgroup and its associated control : face
  * for seborrheic dermatitis of scalp subgroup and its associated control: scalp
  * for telangiectasic erythrocouperosis papule of the face (rosacea) subgroup and its associated control: face
Other: Absorbant paper — * for acne of the face subgroup and its associated control : face
  * for seborrheic dermatitis of scalp subgroup and its associated control: scalp
  * for telangiectasic erythrocouperosis papule of the face (rosacea) subgroup and its associated control: forehead
Other: Hydratation Index — -for atopic dermatitis of the upper limb subgroup and its associated control: upper limb (hand excluded)
Other: TransEpidermal Water Loss — -for atopic dermatitis of the upper limb subgroup and its associated control: upper limb (hand excluded)

SUMMARY:
The physiological states of the skin are characterized by a certain homeostasis linked to the balance of the metabolic pathways. When these pathways are deregulated, the proteic, lipidic and metabolic is affected. It is thus possible to follow a change in the state of the skin by looking at change in the associated molecular profile.

The PRISM laboratory (INSERM U1192) in Lille has developed an innovative system laser called SpiderMass composed of 4 parts:

1. A laser used for the micro-sampling of material in vivo,
2. A transport transfer line of the ablated particles,
3. A mass spectrometer that analyzes them in real time and generates the molecular profiles of the epidermis,
4. A data analysis procedure.

The SpiderMass(TM) is of great interest for the study of the skin because it allows non-invasive vivo characterization, and therefore without biopsy or sample preparation. In addition, it will complement techniques already used in the research center such as FTIR spectroscopy. Indeed, in acne studies the FTIR allows to obtain only the Fatty Acid Triglycerid ratio while the SpiderMass permits to detail these lipid classes by each observed molecule on the surface of the skin and follow their evolution.

ELIGIBILITY:
--> INCLUSION CRITERIA

CRITERIA RELATED TO THE POPULATION:

* Male or female subject having signed a written informed consent for his/her participation to the study
* Subject with a phototype II to IV according to the Fitzpatrick scale
* Subject affiliated to a social security system or health insurance, or is a beneficiary
* For woman of childbearing potential use of an effective method of contraception, as assessed by the investigator for at least 4 weeks before inclusion in the study

For acne of the face subgroup and its associated control: Male or female, 18 to 30 years old included

For atopic dermatitis of the upper limb subgroup and its associated control: Male or female, 20 to 50 years old included

For vulgar plaque psoriasis subgroup and its associated control: Male or female, 20 to 55 years old included

For telangiectasic erythrocouperosis papule of the face (rosacea) subgroup and its associated control: Male or female, 30 to 55 years old included

For seborrheic dermatitis of scalp subgroup and its associated control: Male or female, 20 to 45 years old included

CRITERIA RELATED TO DERMATOSIS:

For subjects of the acne of the face subgroup :

-Subjects with mild to severe acne on the face with a GEA (Global Acne Evaluation) score of 2 to 4 on a rating scale ranging from 0 (no injury) to 5 (very severe)

* Subject presenting on the face, at least one zone:

  * Lesional in immediate border of a papule
  * Peri-lesional near inflammatory lesions (papule, about 1 cm)
* Subject presenting on the inner side of the forearm a reference zone without lesion

For subjects in the atopic dermatitis subgroup of upper limbs:

* Subject with atopic dermatitis on the upper limbs, mild to moderate with SCORAD (SCORing Atopic Dermatitis) between 15 and 40 included with:

  •A dryness score ≥ 2 on a scale ranging from 0 (absent) to 3 (severe)
* Subject having at least one inflammatory flare of atopic dermatitis on the upper limbs in the 2 years before the day of inclusion
* Subject presenting on the upper limb (hand excluded) at least one zone:

  •Lesional defined by the signs of target SCORAD between 3 and 12:

  • Erythema from 1 to 3

  • Dryness ≥2

  • Oedema / papule from 0 to 3
  * Lesions oozing or crusting 0
  * Excoriation of 0
  * Lichenification from 0 to 3 On a scale ranging from 0 (absent) to 3 (severe)
  * Peri-lesional near the lesion zone (about 1cm)
* Subject presenting on the inner side of the forearm a reference zone without lesion

For vulgar plaque psoriasis subgroup

* Subject with mild to moderate erythematous-squamous plaque psoriasis whose IGA (Investigator Global Assessment) score is between 2 and 3, on a rating scale ranging from 0 (clear) to 5 (very severe)
* Subject with on the upper limb (hand excluded) or lower limb at least one zone:

  * Lesional:
  * Without fissure and without crust
  * With erythema score ≥ 1 on a scale ranging from 0 (absent) to 3 (severe)
  * With desquamation score between 1 (mild) and 2 (moderate) on a scale ranging from 0 (absent) to 3 (severe)
  * With an oedema score of 0 (absent) on a scale ranging from 0 (absent) to 3 (severe)
  * Peri-lesional:
  * Without fissure and without crust
  * Near the lesion zone (about 1 cm)
  * Subject presenting on the inner side of the forearm a reference zone without lesion

For telangiectasic erythrocouperosis papule of the face (rosacea) subgroup

- Subject with telangiectasic erythrocouperosis and papule of the face mild to moderate with an IGA score between 2 and 3 on a rating scale ranging from 0 (absent) to 4 (severe)

* Subject presenting on the face at least one zone:

  • Lesional: immediate border of the papule with a persistent erythema score ≥ 1 on a rating scale ranging from 0 (absent) to 3 (severe)

  • Peri-lesional:

  • Near inflammatory lesions (papule, about 1 cm)

  • Ranging of at least 1 point less in the erythema score compared to the lesion zone
* Subject presenting on the inner side of the forearm a reference zone without lesion

For seborrheic dermatitis of scalp subgroup :

* Subject with mild to moderate seborrheic dermatitis with an IGA score between 2 and 3 on a rating scale ranging from 0 (absent) to 4 (severe)
* Subject presenting on the scalp at least one zone:

  * Lesional:
  * with erythema score ≥ 1 on a scale of 0 (absent) to 3 (severe)
  * with clinically visible scales
  * Peri-lesional:Near the lesion zone (about 1 cm)
* Subject presenting on the inner side of the forearm a reference zone without lesion

  * NON INCLUSION CRITERIA

CRITERIA RELATED TO THE POPULATION:

* For woman of childbearing potential: pregnant or breastfeeding
* Subject unable to understand the information given including study procedures (for linguistic or psychiatric reasons) and to give his/her consent in writing
* Subject who, in the judgement of the investigator, is not likely to be compliant with study-related constraints and requirements
* Subject who has forfeited his/her freedom by administrative or legal award or is under guardianship
* Subject who is in a position likely to represent a conflict of interest and/or is a family member of any people involved in the conduct of the study (secretary, nurse, technician…) of the investigational site
* Subject who is currently participating, who plans to participate or who has participated in another clinical study liable to interfere with the study assessments according to the investigator's assessment

CRITERIA RELATED TO DERMATOSIS AND CUTANEOUS CONDITION:

* Subject with premature cutaneous aging linked to a genetic disease
* Subject with solar erythema in at least one zone under study
* Subject with a tattoo, scar or other dermatological sign on at least one study zone that may interfere with the study according to the investigator's assessment
* Subject with autoimmune disease
* Subject with any type of complication on at least one study area (excoriation type, primary, viral, fungal or parasitic bacterial infection, etc.) according to the investigator's assessment

Criteria for control subgroups:

- Subject with a dermatosis or any type of lesion on the zone corresponding to the lesional, peri-lesional zone or reference zone of the associated subgroup dermatosis likely to interfere with the study according to the investigator's assessment

Criteria for chronic inflammatory dermatitis:

For subjects of the acne of the face subgroup:

- Subject with another dermatosis (chronic / acute, inflammatory, infectious, immune) on the face that could interfere with the study according to the investigator's assessment

For subjects in the atopic dermatitis subgroup of upper limbs:

- Subject with another dermatosis (chronic / acute, inflammatory, infectious, immune) on the upper limb (s) to the study likely to interfere with the study according to the investigator's assessment

For vulgar plaque psoriasis subgroup

* Subject with an isolated palmo-plantar form of psoriasis
* Subject with an isolated form of cutaneous psoriasis other than in plaque (in gout, pustular, erythrodermic or inverted elbow creases (psoriasis of the mucous membranes))
* Subject with another dermatosis (chronic / acute, inflammatory, infectious, immune) on the upper limb (s) and/or lower limb(s) to the study likely to interfere with the study according to the investigator's assessment

For telangiectasic erythrocouperosis papule of the face (rosacea) subgroup

- Subject with another dermatosis (chronic / acute, inflammatory, infectious, immune) on the face that could interfere with the study according to the investigator's assessment

For seborrheic dermatitis of scalp subgroup :

* Seborrheic dermatitis under medical treatment
* Subject with another dermatosis (chronic / acute, inflammatory, infectious, immune) on the scalp likely to interfere with the study according to the investigator's assessment (in particular contact eczema or alopecia)

CRITERIA RELATED TO TREATMENTS AND PRODUCTS

For all subjects :

* Oral intake of isotretinoin or acitretin (oral vit-A and derivatives) within the 6 months prior to the inclusion visit or the day of the visit
* Local retinoid treatment on at least one study zone, which may interfere with the results of the study according to the investigator's assessment within the month preceding the inclusion visit or the day of the visit
* Phototherapy treatment in at least one study zone within 4 weeks prior to the inclusion visit or the day of the visit
* Topical or oral treatment established or modified during the previous weeks or to be established or modified during the study, which may interfere with the results of the study according to the investigator's assessment ( for example modifying the cutaneous characteristics: treatment inducing pigmentation), keratolysis, ...)
* Anti-inflammatory treatment (steroidal or nonsteroidal) taken daily and repeatedly for more than 5 consecutive days during the week preceding the inclusion visit
* Application of any topical vitamin D-derived treatment on at least one study zone within 3 weeks prior to the inclusion visit or the day of the visit
* Application of dermocorticoid topical or immunomodulatory topical treatments (tacrolimus), antifungals, local antibiotics on at least one study zone in the 3 weeks prior to the inclusion visit or the day of the visit
* Application of water, product or topical treatment on at least one zone under study after the last wash the day before the visit
* Application of water, topical product or make-up on at least one zone the day of the inclusion visit

For seborrheic dermatitis of scalp subgroup and its associated control :

* Use on the scalp of any product that can be active on squamous conditions, rinsed or posed (anti-dandruff, anti-fungal shampoo, vinegar rinse, essential oils ...) within 2 weeks prior to the inclusion visit or the day of the visit
* Any technique to change the color or condition of the hair (coloring, discoloration, permanent, smoothing / straightening, ..) performed within 2 weeks prior to the inclusion visit or the day of the visit
* Washing of the scalp done within 2 days before the inclusion visit or the day of the visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Signals and molecular profiles (including lipid) of the epidermis | baseline
  Defined by characteristic peak mass intensities - SpiderMass
Molecular profiles (including lipid) of the epidermis according to sampling method and the measurements of the signals obtained method | baseline
  * sampling method - absorbant paper, in vivo and / or by scotch
  * measurements of the signals obtained -in vivo or FTIR
Cutaneous hydratation for atopic dermatitis subgroup and its associated control | baseline
  By hydratation index - Corneometer
State of the cutaneous barrier for atopic dermatitis and corresponding control volunteers | baseline
  Rate of the Trans Epithelial Water Loss (TEWL) by arbitrary units with an Aquaflux system (Biox Systems Ltd, London. UK)
Global lipid quantity measured on face acnea, scalp seborrheic dermatitis, face rosacea (papulotelangiectasic stage of erythrocouperosis) and corresponding control volunteers | baseline
  Global sebum level measurement expressed in arbitrary index with a Sebumeter SM815 system (Courage+Khazaka electronic GmbH, Köln. Germany)
Skin state evaluation on the lesional and perilesional areas | baseline
  Illustrative descriptions of the skin state with photographs, taken by an iPhone 6S (Apple, Cupertino. Califronia, USA) dedicated to the study
Impact of several factors (dermatosis, area, gender, age) on the molecular profiles of the epidermis | baseline
  Characteristic peak mass intensities - SpiderMass

CONTACTS AND LOCATIONS:
Overall Officials: Thérèse NOCERA, Mrs, Principal Investigator — Centre de Recherche sur La Peau
Locations (1):
- Centre de Recherche sur la Peau, Toulouse, France